CLINICAL TRIAL: NCT06689033
Title: Comparison of High Flow Nasal Oxygen and Standard Nasal Oxygen in Preventing Hypoxia in Patients Undergoing Endoscopic Retrograde Cholangiopancreatography Under Sedation
Brief Title: High Flow Nasal Oxygen Versus Standard Nasal Oxygen in Endoscopic Retrograde Cholangiopancreatography Under Sedation
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Other Study IDs: E2-23-4070
Record Dates: First submitted 2024-10-28; First posted 2024-11-14 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde; Hypoxia; Sedation
Keywords: HFNO; sedation; prone position; Cholangiopancreatography, Endoscopic Retrograde
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Group 1: Patients sedated for ERCP, receiving nasal oxygen: Nasal Oxygen, preoxygenation with 100% oxygen for 3 min with an oxygen flow rate of 8 L.min-1 via a nasal cannula before induction and 100% oxygen with a flow rate of 5 L.min-1 throughout the procedure.
- Group 2: Patients sedated for ERCP receiving high flow nasal oxygen: High flow nasal oxygen, preoxygenation with 100% oxygen with a flow rate of 40 L.min-1 for 3 min before induction and received 50% oxygen with a flow rate of 50 L.min-1.

SUMMARY:
The administration of supplemental oxygen using a standard nasal cannula is the current standard of care for patients undergoing sedation for gastrointestinal endoscopic procedures. Endoscopic Retrograde Cholangio Pancreatography can be particularly challenging for anesthesiologists due to the increased difficulty in airway access when performed in the prone position. High-flow nasal oxygen is a non-invasive oxygen therapy system that can provide heated and humidified air containing oxygen at a high flow rate.This study aims to compare the effectiveness of High Flow Nasal Oxygen versus standard nasal oxygen in preventing hypoxemia in patients undergoing deep sedation during ERCP procedures.

DETAILED DESCRIPTION:
Ankara City Hospital's Gastrointestinal Endoscopy Colonoscopy Unit's patient count determined using G-power statistical software ensured that a sample size of at least 185 patients was adequate at a 95% confidence level with 80% power and an effect size of 0.5. Analyses were performed using the Power and Sample Size statistical program version 3.1.2 (Vanderbilt University, 2015).

187 patients scheduled for ERCP procedure under sedation during an 8-month period were included in the study. The study was planned as a randomized observational and prospective study. Patients were randomly allocated to either the nasal oxygen (NO) or High Flow Nasal Oxygen (HFNO) group in a 1:1 ratio using a computer-generated random code generator. It was not a blind study, as the oxygen delivery systems did not look the same. Endoscopists, anesthesiologists, and patients were not blinded. ERCP procedures were completed by one of two expert endoscopists and sedation was performed by one of two anesthesiologists trained in endoscopic sedation. The study and possible risks were explained to all patients participating in the study, and written informed consent was obtained from the patients. The patient's age, current chronic diseases, and duration of the procedure were recorded. Before the procedure, the frailty level of the patients was evaluated with the Modified Frailty Index-11 (mFI-11) and recorded. The mFI-11 is an 11-item index that assesses comorbidities to stratify patient risk. The simplified frailty index is calculated as the number of present comorbidities divided by the total number of 11 items used in the mFI-11 assessment, which includes diabetes mellitus, not independent functional status, chronic obstructive pulmonary disease, congestive heart failure, myocardial infarction, percutaneous coronary intervention or cardiac surgery, angina, hypertension medication, peripheral vascular disease, impaired sensorium, transient ischemic attack, and cerebrovascular accident. The resulting score ranges from 0 to 1. Patients were positioned prone and pulse oximetry, non-invasive blood pressure monitoring, electrocardiography, and Bispectral Index monitoring were performed, and baseline values were recorded in all cases. The NO group was preoxygenated with 100% oxygen for 3 min with an oxygen flow rate of 8 L.min-1 via a nasal cannula before induction and received 100% oxygen with a flow rate of 5 L.min-1 throughout the procedure. The HFNO group was preoxygenated with 100% oxygen with a flow rate of 40 L.min-1 for 3 min via an HFNO system (Inspired 02FLO High Flow Heated Respiratory Humidifier, VUN-001, Vincent Medical Manufacturing Co., Hong Kong) before induction and received 50% oxygen with a flow rate of 50 L.min-1. In case of a decrease in saturation (SpO2<90), the flow was increased to 60 L.min-1, and if it did not resolve, FiO2 was increased to 100%. All patients were premedicated with iv midazolam and sedation was performed with iv 1 µg.kg-1 fentanyl and iv bolus dose of 0.5-1 mg.kg-1 %1 propofol followed by an iv infusion of propofol 3-4 mg.kg-1.hr-1 targeting a BIS value of 60-80. In case of apnea or desaturation, maneuvers such as patient stimulation, chin lifting, or increasing oxygen flow were performed and recorded. The lowest SpO2 values obtained for both groups were noted.

The data were analyzed using IBM SPSS Statistics ver. 25 (IBM Corporation, Armonk, NY, USA). The distribution of continuous numerical variables was tested for normality using the Kolmogorov-Smirnov test, and the homogeneity of variances was assessed with Levene's test. Descriptive statistics were expressed as mean ± standard deviation or range (minimum - maximum) for continuous variables, and as case number and percentage (%) for categorical variables. The significance of differences between the NO and HFNO groups for continuous variables that met the assumptions of parametric test statistics was evaluated using Student's t-test, whereas differences for those that did not meet these assumptions were assessed using the Mann-Whitney U test. The significance of changes over time in systolic, diastolic, and mean blood pressure, heart rate, oxygen saturation (SpO2), and BIS levels was examined using repeated measures analysis of variance with Wilks' Lambda test. Where Wilks' Lambda test results were found significant, the specific times causing the differences were identified using the Bonferroni-adjusted multiple comparison test. Comparisons between the NO and HFNO groups were made by calculating the changes in SpO2 and BIS from baseline at subsequent time points. Unless otherwise stated, Pearson's χ2 test was used for the analysis of categorical data. For 2x2 contingency tables where at least 25% of the expected frequencies were below 5, Fisher's exact test was used, and where expected frequencies were between 5 and 25, the continuity-adjusted χ2 test was employed. In RxC tables (where at least one of the categorical variables in the row or column had more than two outcomes), if at least 25% of the cells had expected frequencies below 5, the Fisher-Freeman-Halton test was applied. Unless stated otherwise, results were considered statistically significant at p<0.05. However, to control for Type I error in all multiple comparisons, Bonferroni correction was applied.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary patients over 18 years of age
* ASA (American Society of Anaesthesiologists) I-IV risk scores

Exclusion Criteria:

* Patients with altered mental status, dementia, cognitive disorders
* Intubation
* Tracheostomies
* Need for oxygen therapy due to preexisting disease
* Pregnancy
* Recent history of nasal bleeding
* Allergy to propofol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for ERCP procedure under sedation in Ankara City Hospital's Gastrointestinal Endoscopy Colonoscopy Unit are included.
Sampling Method: Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Oxygen saturation SpO2 levels of the cases in % | Oxygen saturation levels were recorded before induction and every 5 minutes throughout the procedure that lasted around 30 minutes.
  Each patient was monitored with an oxygen saturation probe and SpO2 levels of the cases were recorded before induction of sedation and every 5 minutes, throughout the procedure. Hypoxemia was detected.

SECONDARY OUTCOMES:
Number of interventions over procedure time (number) | Number of maneuvers performed throughout the procedure, that lasted around 30 minutes were recorded.
  In case of apnea or desaturation, airway interventions were performed and recorded throughout the procedure

OTHER OUTCOMES:
Systolic, diastolic and mean blood pressures were recorded | Blood pressure monitorization was performed before induction and every 5 minutes throughout the procedure that lasted around 30 minutes.
  Before induction patients were monitored, and systolic, diastolic and mean blood pressures were recorded before induction and every 5 minutes throughout the procedure.
Heart beat was recorded in beats per minute | Heart beat monitorization was performed before induction and every 5 minutes throughout the procedure that lasted around 30 minutes.
  Heart beats were recorded before induction and every 5 minutes throughout the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Ezgi Erkilic, Associate Professor, Principal Investigator — Ankara Bilkent City Hospital, Department of Anesthesiology
Locations (1):
- Ankara Bilkent City Hospital, Department of Anesthesiology, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after publication of the study. Study protocol, statistical analysis, study report will be shared if required by a researcher.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning right after publication and ending 2 years after the publication of results
Access Criteria: Data required for research and meta-analysis will be shared.

REFERENCES:
- [Background] Carron M, Tamburini E, Safaee Fakhr B, De Cassai A, Linassi F, Navalesi P. High-flow nasal oxygenation during gastrointestinal endoscopy. Systematic review and meta-analysis. BJA Open. 2022 Oct 18;4:100098. doi: 10.1016/j.bjao.2022.100098. eCollection 2022 Dec. PMID 37588780
- [Background] Sawase H, Ozawa E, Yano H, Ichinomiya T, Yano R, Miyaaki H, Komatsu N, Ayuse T, Kurata S, Sato S, Pinkham MI, Tatkov S, Ashizawa K, Nagata K, Nakao K. Respiratory support with nasal high flow without supplemental oxygen in patients undergoing endoscopic retrograde cholangiopancreatography under moderate sedation: a prospective, randomized, single-center clinical trial. BMC Anesthesiol. 2023 May 8;23(1):156. doi: 10.1186/s12871-023-02125-w. PMID 37158818
- [Background] Zhang YX, He XX, Chen YP, Yang S. The effectiveness of high-flow nasal cannula during sedated digestive endoscopy: a systematic review and meta-analysis. Eur J Med Res. 2022 Feb 24;27(1):30. doi: 10.1186/s40001-022-00661-8. PMID 35209948
- [Background] Douglas N, Ng I, Nazeem F, Lee K, Mezzavia P, Krieser R, Steinfort D, Irving L, Segal R. A randomised controlled trial comparing high-flow nasal oxygen with standard management for conscious sedation during bronchoscopy. Anaesthesia. 2018 Feb;73(2):169-176. doi: 10.1111/anae.14156. Epub 2017 Nov 24. PMID 29171661
- [Background] Corral-Blanco M, Sayas-Catalan J, Hernandez-Voth A, Rey-Terron L, Villena-Garrido V. High-Flow Nasal Cannula Therapy as an Adjuvant Therapy for Respiratory Support during Endoscopic Techniques: A Narrative Review. J Clin Med. 2023 Dec 22;13(1):81. doi: 10.3390/jcm13010081. PMID 38202089
- [Background] Cha B, Lee MJ, Park JS, Jeong S, Lee DH, Park TG. Clinical efficacy of high-flow nasal oxygen in patients undergoing ERCP under sedation. Sci Rep. 2021 Jan 11;11(1):350. doi: 10.1038/s41598-020-79798-7. PMID 33432035
- [Background] Lee MJ, Cha B, Park JS, Kim JS, Cho SY, Han JH, Park MH, Yang C, Jeong S. Impact of High-Flow Nasal Cannula Oxygenation on the Prevention of Hypoxia During Endoscopic Retrograde Cholangiopancreatography in Elderly Patients: A Randomized Clinical Trial. Dig Dis Sci. 2022 Aug;67(8):4154-4160. doi: 10.1007/s10620-021-07272-z. Epub 2021 Nov 2. PMID 34727281
- [Background] Kim SH, Bang S, Lee KY, Park SW, Park JY, Lee HS, Oh H, Oh YJ. Comparison of high flow nasal oxygen and conventional nasal cannula during gastrointestinal endoscopic sedation in the prone position: a randomized trial. Can J Anaesth. 2021 Apr;68(4):460-466. doi: 10.1007/s12630-020-01883-2. Epub 2021 Jan 6. PMID 33403549